CLINICAL TRIAL: NCT05288764
Title: Correlation Between Concentration at the Effector Site of Ketamine (Calculated With DOMINO Pump) and Bispectral Index Values During General Anaesthesia for Breast Surgery.
Brief Title: Effect of Ketamine on BIS Values
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, University of Padova
Other Study IDs: KetaMAST
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia Brain Monitoring; Ketamine
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bispectral Index — Comparing Bispectral index values (usually adopted during general anaesthesia monitoring) to Ketamine concenetration at the effector site calculated with Domino model pump (usually adopted for Ketamine infusion during general anaesthesia)

SUMMARY:
Aim of this trial is to define if Concentration at the effector site (Ce) of Ketamine, calculated with DOMINO model infusion pump are correlated with Bispectral Index BIS values during general anaesthesia for breast surgery.

DETAILED DESCRIPTION:
Correlation between Concentration at the effector site (Ce) of Ketamine and Bispectral Index (BIS) values during general anaesthesia for breast surgery has not been defined yet.

We want to analyze this correlation during general anaesthesia conducted using Propofol, ketamine and remifentanil. All of these drugs will be delivered with Targeted-ControlledInfusion pumps (in particular Eleveld for Propofol, Minto for Remifentanil and Domino for Ketamine).

ELIGIBILITY:
Inclusion Criteria:

* Undergo gneral anaesthsia with Targted Controlld Infusion of Ketamine (Domino model), Propofol (Schnider model) and Remifentanil (Minto model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Benzodiazepiones absuntion
* Obesity

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing brast cancer surgery
Study Population: Adult Women undergoing breast surgery for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Concentration at the effector site of Ketamine and BIS values | We will collected data about Drugs concentration and BIS values during general anaesthesia. We will collect BIS and TCI Ketamine values during all the duration of anesthesia, form the start of ketamine bolus until the emergence from anesthesia
  Discover if there is linear correlation between Concentration at the effector site of Ketamine and BIS values during standard general anaesthesia conducted with Propofol, remifenatnil and ketamine delivered with targeted controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS 2 Marca Trevigiana, Treviso, Tv, Italy

REFERENCES:
- [Derived] Linassi F, Troyas C, Kreuzer M, Spano L, Burelli P, Schneider G, Zanatta P, Carron M. Effect of Ketamine on the Bispectral Index, Spectral Edge Frequency, and Surgical Pleth Index During Propofol-Remifentanil Anesthesia: An Observational Prospective Trial. Anesth Analg. 2025 Jun 1;140(6):1276-1285. doi: 10.1213/ANE.0000000000007255. Epub 2024 Nov 1. PMID 39485729